CLINICAL TRIAL: NCT04697498
Title: Bilateral Bi-level Erector Spine Plane Block as a Component of General Anesthesia in Surgical Correction of Spinal Deformations
Acronym: BBESPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Maksym Barsa, Principal Investigator, Lviv National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNMY-FPGE- ANESTHESIOLOGY-BBES
Record Dates: First submitted 2020-12-29; First posted 2021-01-06 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Scoliosis; Spinal Deformity; Acute Pain; Chronic Pain; Postoperative Pain; Anesthesia; Regional Anesthesia Morbidity; Anesthesia, Local; Anesthesia Complication; Hyperalgesia; Intraoperative Complications; Intraoperative Hypotension; Intraoperative Blood Loss; Intraoperative Bleeding; Intraoperative Neurological Injury; Intraoperative Injury; Coagulation Disorder; Postoperative Nausea and Vomiting; Postoperative Cognitive Dysfunction; Neuropathic Pain; Nutrient Deficiency; Nutrition Disorders; Ventilator-Induced Lung Injury
Keywords: Erector spinae plane block; Regional anesthesia; Scoliosis; Spinal Deformity; Multimodal analgesia
MeSH Terms: conditions — Scoliosis; Acute Pain; Chronic Pain; Pain, Postoperative; Hyperalgesia; Intraoperative Complications; Blood Loss, Surgical; Hemostatic Disorders; Postoperative Nausea and Vomiting; Postoperative Cognitive Complications; Neuralgia; Nutrition Disorders; Ventilator-Induced Lung Injury | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Control Group (Active Comparator): The control group will include patients who will undergo surgery under general anesthesia.
  Interventions: Procedure: General anaesthesia
- The Study Group (Experimental): The study group will include patients who will undergo surgery under general anesthesia using a bilateral bi-level Erector spine plane block.
  Interventions: Procedure: Bilateral bi-level Erector spine plane block

INTERVENTIONS:
Procedure: Bilateral bi-level Erector spine plane block — After intubation of the trachea and rotation on the abdomen before the skin incision will be performed bilateral bi-level Erector spine plane block. Before surgery, the level of screw placement will be discussed with the surgeon, and the blockade will be performed at two levels of the spine bilaterally as close as possible to the screw placement site. For blockade a solution for prolonged blockade of peripheral nerve plexuses with bupivacaine 0.375%, dexamethasone 0.02% and epinephrine 0.00018% will be used.
  Arms: The Study Group
Procedure: General anaesthesia — The control group - will include patients who will undergo surgery under general anaesthesia
  Arms: The Control Group

SUMMARY:
Improving the anesthesiology management for surgical correction of spinal deformations with introducing the diagnostic methods and treatment strategy of acute pain, preventing the evolution of chronic pain. Development and implementation in clinical practice perioperative intensive care protocols for surgical correction of spinal deformities.

DETAILED DESCRIPTION:
The study will involve patients for whom are indicated a surgical correction of spinal deformations.

The control group will include patients who will undergo surgery under general anesthesia. The study group will include patients who will undergo surgery under general anesthesia using a bilateral bi-level Erector spine plane block.

Stages of the study: preoperative period, onset of anesthesia (induction of anesthesia), maintenance of anesthesia, end of anesthesia, 6th and 12th hours after surgery, 1st, 3rd, 5th day after surgery.

All patients will be given the same preparation for surgery: 5-7 days before the procedure - erythropoietin (50-75 IU / kg) subcutaneously once; iron 100 mg iv daily; thiamine hydrochloride (50 mg), pyridoxine hydrochloride (50 mg), cyanocobalamin (0.5 mg) and ascorbic acid (500 mg) orally, daily. The condition of the cardiovascular and respiratory systems will be assessed by auscultation and percussion of the heart and lungs, the results of electrocardiography, echocardiography, spirometry will by also estimate, vascular Doppler of the lower extremities and neck will by also performed.

Blood tests will be taken before and after surgery (haemoglobin, erythrocytes, leukocytes, colour index, haematocrit, leukocyte formula, erythrocyte sedimentation rate, blood glucose, coagulogram, electrolytes, creatinine, urea, albumin, bilirubin, transaminases, cortisol, testosterone, c-reactive protein).

Patients will be given recommendations on proper nutrition before surgery (solid food is allowed 6 hours before surgery and 150 ml of sweet clear liquid 2 hours before surgery), hospitalization will take place on the day of surgery.

All patients will have two peripheral veins cannulated and a urethral catheter will be installed before surgery. In patients with scoliotic spinal deformity, a central venous catheter will be inserted into the right jugular vein under ultrasound guidance prior to surgery. Antibiotic prophylaxis will be performed two hours before the skin incision. Mechanical bowel preparation and premedication with sedatives will not be performed.

All patients in the operating room will receive paracetamol, dexketoprofen, ondansetron, diphenhydramine, dexamethasone, atropine, tranexamic acid. For induction of anesthesia - propofol, thiopental, fentanyl, atracurium besylate, suxamethonium iodide. After preoxygenation - intubation of the trachea in an improved position and further rotation on the abdomen with specific placement of the patient to prevent compression of the abdominal cavity. In patients with scoliotic spinal deformity in the abdominal position will be used a lung recruitment manoeuvre (gradual increasing in positive end-expiratory pressure and inspiratory pressure with assessment of tidal volume and lung pliability), and subsequent protective ventilation and supporting Driving Pressure 12-14 cm H2O.

The operation will be performed under general inhalation anesthesia with sevoflurane and dexmedetomidine infusion. In patients undergoing neuromonitoring, relaxants will be administered only for tracheal intubation.

Intraoperatively, all patients will be monitored for electrocardiography, respiratory rate, body temperature, systolic, diastolic and mean blood pressure, heart rate, pulse oximetry.

During the operation, an assessment of blood loss and subsequent balanced infusion therapy will be performed. The volume and rate of urination will be assessed. A constant infusion of tranexamic acid will be established. Controlled arterial hypotension with mean blood pressure of at least 60 mm Hg will be maintained. To protect the spinal cord and its roots from ischemic injury during the derotation maneuver, mean blood pressure will be maintained at normal or elevated levels.

Correction of blood loss will be carried out with balanced solutions of crystalloids. Blood transfusion will be started at Hb less than 90 g / l. Patients will be warmed by the Warm Touch heating system. All patients will be extubated in the early postoperative period.

For the purpose of analgesia in the postoperative period, patients of both groups will receive paracetamol and dexketoprofen, thromboprophylaxis will be performed depending on the risk of thromboembolic complications.

In the study group, after intubation of the trachea and rotation on the abdomen before the skin incision will be performed bilateral bi-level Erector spine plane block. Before surgery, the level of screw placement will be discussed with the surgeon, and the blockade will be performed at two levels of the spine bilaterally as close as possible to the screw placement site. For blockade a solution for prolonged blockade of peripheral nerve plexuses with bupivacaine 0.375%, dexamethasone 0.02% and epinephrine 0.00018% will be used (Patent №133643 Ukraine 'Solution for prolonged blockade of peripheral nerve plexuses' inventor and owner Barsa Maksym № u201900272, declared 10.01.2019, valid from 10.04.2019, Bulletin № 7).

The total amount of solution administered is 40 ml (10 ml per injection). The erector spine muscle and the transverse process of the spine will be identified using a linear ultrasound probe at the required level of the spine 3cm laterally from the spinous process. Then, using an echogenic needle under ultrasound control in a space between the Erector spine muscle and the transverse process bilaterally on two levels of the spine a local anaesthetic with adjuvants will be injected (Patent №140510 Ukraine 'Method of anaesthesiologic securement for surgical correction of scoliosis spinal deformity' inventor and owner Barsa Marsym № u201911515, claimed 28.11.2019, valid from 25.02.2020, Bulletin № 4).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of the patient or his legal representatives to participate the study.
2. Spinal deformity that requires surgical correction.
3. No known allergies to local anaesthetics.
4. Negative intradermal test for sensitivity to local anaesthetics.

Exclusion Criteria:

1. Refusal of the patient or his legal representatives to participate the study
2. Diabetes mellitus, known allergy to local anaesthetics
3. Acute spinal cord injury
4. Physical status according to classification ASA III and more
5. A positive intradermal test for sensitivity to a local anaesthetic.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in The Numeric Pain Rating Scale | On the 1st, 2rd and 3th day after surgery
  The 11-point numeric scale ranges from '0' representing one pain extreme - "no pain"; to '10' representing the other pain extreme - "pain as bad as you can imagine" or "worst pain imaginable". Will be measured in rest and in the movement.
Duration of hospitalization | Through study completion, an average of 1 year
Time of weaning the patient from mechanical ventilation | From a few minutes to an hour

SECONDARY OUTCOMES:
The amount of opioid administered during surgery and in the postoperative period | Through study completion, an average of 1 year
Mechanical pain threshold and sensitivity | Baseline, on the 1st, 3rd and 5th day after surgery
  A set of 20 calibrated von Frey monofilaments will be used to determine the mechanical pain threshold. We will make pressure by the monofilament on the skin with increasing force from 0.008 grams to 180 grams. The patient will be asked to close his eyes and we will press the monofilament to the skin surface at an angle of 90 ° until the monofilament bends for 1-1.5 seconds. Monofilaments will be used in ascending order. An interval of 10 s will be maintained between studies. Mechanical pain threshold will be defined as the lowest force of pressure that will be perceived by the patient as pain. Determination of the mechanical pain threshold will be performed in two areas - on the palmar surface of the forearm and on the scapular lines.
Overall satisfaction with analgesia will be assessed on a 5-point Likert scale | Through study completion, an average of 1 year
  A type of psychometric response scale in which responders specify their level of satisfaction with analgesia in five points: 5 - Excellent, 4 - Good, 3 - More or less good (pretty good), 2 - Bad, 1 - Very bad.
Level of postoperative sedation will be assessed with Richmond Agitation-Sedation Scale | On the 1st day after surgery
  A medical scale used to measure the agitation or sedation level of a person. (+4) - Combative (Overtly combative or violent; immediate danger to staff); (+3) - Very agitated (Pulls on or removes tubes or catheters or has aggressive behavior toward staff); (+2) - Agitated (Frequent nonpurposeful movement or patient-ventilator dyssynchrony); (+1) - Restless (Anxious or apprehensive but movements not aggressive or vigorous); (0) - Alert and calm (Spontaneously pays attention to caregiver); (-1) - Drowsy (Not fully alert, but has sustained, more than 10 seconds, awakening, with eye contact, to voice); (-2) - Light sedation (Briefly, less than 10 seconds, awakens with eye contact to voice); (-3) - Moderate sedation (Any movement, but no eye contact, to voice); (-4) - Deep sedation (No response to voice, but any movement to physical stimulation); (-5) - Unarousable (No response to voice or physical stimulation)
In the group of patients which will undergo general anaesthesia with Erector spine plane block, anaesthetised dermatomes will be counted along the paravertebral, scapular, anterior, middle and posterior axillary, midclavicular and parasternal lines | Baseline, 1st day after surgery
  It will be measured by response to von Frey hair stimulation
Blood glucose level | Baseline, 1st and 5th day after surgery
Blood testosterone level | Baseline, 1st and 5th day after surgery
Blood cortisol level | Baseline, 1st and 5th day after surgery
Blood C-reactive protein level | Baseline, 1st and 5th day after surgery
Erythrocyte sedimentation rate | Baseline, 1st and 5th day after surgery
Mean blood pressure | Baseline, during and 1st hour after surgery
Heart rate | Baseline, during and 1st hour after surgery
Nociceptive respond index | Every 15 minutes during surgery
  The nociceptive response index was calculated every 15 minutes during surgery, using the nociceptive response index formula, which includes the intra-operative haemodynamic variables HR, SBP and perfusion index
Blood loss | Baseline, during and 1st hour after surgery
  By weighing the wipes before and after use, measuring the amount of blood in the suction flask.
Urination | Baseline, during and 1st hour after surgery
Infusion therapy | Baseline, during and 1st hour after surgery
Episodes of nausea, belching, vomiting and constipation | Five days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maksym Barsa, Principal Investigator — Rivne Region Hospital
Locations (1):
- Rivne Oblast State Hospital, Rivne, Rivne Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.22141/2224-0586.16.6.2020.216516